CLINICAL TRIAL: NCT04788563
Title: Heat-sensitive Moxibustion Self-administration for Primary Hypertension in Community: A Multicenter, Pragmatic, Randomized Controlled Trial With Patient Preference Arms
Brief Title: A Randomized Patient Preference Trial on Heat-sensitive Moxibustion for Primary Hypertension in Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhou, Associate professor, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JXUTCM-Mox-02
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with patient preference arms
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Heat-sensitive moxibustion group A (Experimental): In this group, patients are compulsively randomized to receive heat-sensitive moxibustion. They will maintain their original antihypertensive treatment (antihypertensive drugs or no treatment).
  Interventions: Other: Heat-sensitive moxibustion plus original antihypertensive treatment (compulsively randomized arm)
- Control group A (Active Comparator): In this group, patients are compulsively randomized to not receive heat-sensitive moxibustion. They will maintain their original antihypertensive treatment (antihypertensive drugs or no treatment).
  Interventions: Drug: Original antihypertensive treatment (compulsively randomized arm)
- Heat-sensitive moxibustion group B (Experimental): Patients who voluntarily choose to receive randomization and are randomly assigned to receive heat-sensitive moxibustion. They will maintain their original antihypertensive treatment (antihypertensive drugs or no treatment).
  Interventions: Other: Heat-sensitive moxibustion plus antihypertensive treatment (voluntarily randomized arm)
- Control group B (Active Comparator): Patients who voluntarily choose to receive randomization and are randomly assigned to not receive heat-sensitive moxibustion. They will maintain their original antihypertensive treatment (antihypertensive drugs or no treatment).
  Interventions: Drug: Original antihypertensive treatment (voluntarily randomized arm)
- Heat-sensitive moxibustion group C (Experimental): Patients who voluntarily choose to receive heat-sensitive moxibustion. They will maintain their original antihypertensive treatment (antihypertensive drugs or no treatment).
  Interventions: Other: Heat-sensitive moxibustion plus original antihypertensive treatment (preference selection arm)
- Control group C (Active Comparator): Patients who voluntarily choose to not receive heat-sensitive moxibustion. They will maintain their original antihypertensive treatment (antihypertensive drugs or no treatment).
  Interventions: Drug: Original antihypertensive treatment (preference selection arm)

INTERVENTIONS:
Other: Heat-sensitive moxibustion plus original antihypertensive treatment (compulsively randomized arm) — In this group, patients will self-administer heat-sensitive moxibustion or have family members help with the administration for six months. During this period, they will maintain their original antihypertensive treatment.
  Arms: Heat-sensitive moxibustion group A
Drug: Original antihypertensive treatment (compulsively randomized arm) — In this group, patients will maintain their original antihypertensive treatment.
  Arms: Control group A
Other: Heat-sensitive moxibustion plus antihypertensive treatment (voluntarily randomized arm) — In this group, patients will self-administer heat-sensitive moxibustion or have family members help with the administration for six months. During this period, they will maintain their original antihypertensive treatment.
  Arms: Heat-sensitive moxibustion group B
Drug: Original antihypertensive treatment (voluntarily randomized arm) — In this group, patients will maintain their original antihypertensive treatment.
  Arms: Control group B
Other: Heat-sensitive moxibustion plus original antihypertensive treatment (preference selection arm) — In this group, patients will self-administer heat-sensitive moxibustion or have family members help with the administration for six months. During this period, they will maintain their original antihypertensive treatment.
  Arms: Heat-sensitive moxibustion group C
Drug: Original antihypertensive treatment (preference selection arm) — In this group, patients will maintain their original antihypertensive treatment.
  Arms: Control group C

SUMMARY:
Heat-sensitive moxibustion, an important mean of external therapy of traditional Chinese medicine, has unique advantages in treating various chronic diseases than common moxibustion. This study aims to evaluate the efficacy, safety, and cost-effectiveness of heat-sensitive moxibustion for primary hypertension under community self-management setting using a multicenter, pragmatic, randomized controlled trial design with patient-preference arms.

DETAILED DESCRIPTION:
Primary hypertension is a common chronic disease that threatens the life and health of human beings. The conventional western drug therapy often has side effects and many patients are unable to achieve ideal blood pressure control with drugs alone. Therefore, the treatment of primary hypertension still requires active exploration of complementary and alternative therapies with clear clinical efficacy.

Heat-sensitive moxibustion is an innovative moxibustion therapy. By stimulating the patient's special moxibustion sensation, heat-sensitive moxibustion can achieve better results than traditional moxibustion for many diseases, including primary hypertension. Heat-sensitive moxibustion is an easy, inexpensive and safe treatment method. The practitioner does not need to be professionally qualified to perform moxibustion, making it a suitable technique for patients to self-medicate on a daily basis. Traditional moxibustion has been shown to lower blood pressure in patients with primary hypertension. Theoretically, heat-sensitive moxibustion could achieve better blood pressure lowering effects, but its effects in lowering blood pressure in the setting of self-management in community patients is unclear. To verify the efficacy and safety of heat-sensitive moxibustion community self-management for hypertension, we plan to perform a randomized controlled trial. In this trial, we designed the trial grouping scheme as a randomized controlled trial with patient preference arms in order to improve patient adherence and reduce the impact of patient preference effects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with essential hypertension, i.e., systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90 mmHg, with a course more than 6 months.
2. Ages: 18-80 years;
3. The original antihypertensive drugs are calcium channel blockers and/or angiotensin II receptor blockers.
4. Did not receive acupoint stimulation therapies for hypertension in the last month.
5. Patients in the heat-sensitive moxibustion groups need to develop at least one type of moxibustion sensation around the following acupoints: Yongquan, Baihui, Shenque, Quchi, Zusanli, Hegu, Taichong and Dazhui.
6. Consent to sign an informed consent form

Exclusion Criteria:

1. Systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥ 110mmHg after taking antihypertensive drugs;
2. Secondary hypertension.
3. Pregnancy and lactation;
4. Allergic to moxibustion devices, moxa smoke or Artemisia argyi.
5. Complicated with severe diseases that are not recommended for heat-sensitive moxibustion, such as acute cerebral hemorrhage, hypertensive crisis, sensory disturbances, serious mental diseases, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline and months 1, 2, 3, 4, 5, and 6
  Changes from baseline in systolic blood pressure

SECONDARY OUTCOMES:
Diastolic blood pressure | Baseline and months 1, 2, 3, 4, 5, and 6
  Changes from baseline in diastolic blood pressure
Response to treatment | Baseline and months 1, 2, 3, 4, 5, and 6
  Definition: (i) a decrease in systolic blood pressure ≥ 20 mmHg or diastolic blood pressure ≥ 10 mmHg; or (ii) blood pressure control of < 140 mmHg systolic and < 90 mmHg diastolic in patients aged ≥ 65 years; blood pressure control of < 130 mmHg systolic and < 80 mmHg diastolic in patients aged < 65 years.
Dose of antihypertensive drugs | Measure at baseline screening, monthly for 6 months
  Changes from baseline in dose of antihypertensive drugs
Score of EQ-5D-5L | Baseline and months 3 and 6
  Quality of life will be measured using Euro-Qol-5 Dimensions-5 Levels questionnaire (EQ-5D-5L)
Symptom score | Baseline and months 3 and 6
  Symptoms will be scored using the scale in "Guiding Principles of Clinical Research on New Drugs of Chinese Medicines"
Cost-effectiveness ratio | Baseline and months 1, 2, 3, 4, 5, and 6
  Outpatient and inpatient costs for each group will be recorded and used to calculate the cost-effectiveness ratio
Patients' compliance to heat-sensitive moxibustion | Baseline and months 1, 2, 3, 4, 5, and 6
  Patients' compliance will be assessed by recording the frequency and duration of heat-sensitive moxibustion.
Incidence of cardiovascular events | Baseline and months 1, 2, 3, 4, 5, and 6
  Newly developed cardiovascular events
Any adverse events | Baseline and months 1, 2, 3, 4, 5, and 6
  Adverse event data will be derived from patient self-reports and physician reviews.
Heat-sensitive moxibustion-related adverse events | Baseline and months 1, 2, 3, 4, 5, and 6
  Heat-sensitive moxibustion-related adverse event data will be derived from patient self-reports and physician reviews.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhou, M.D., Principal Investigator — Jiangxi University of Traditional Chinese Medicine
Locations (7):
- China (7):
  - Erliuling, Nanchang, Jiangxi
  - Hongmiao, Nanchang, Jiangxi
  - Jinghexinggong community, Nanchang, Jiangxi
  - Jinsheng community, Nanchang, Jiangxi
  - Nangang community, Nanchang, Jiangxi
  - Shajing, Nanchang, Jiangxi
  - Wuliangdian community, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou X, Li S, Li L, Deng G, Dai L, Chai L, Wu Q, Yao Z, Deng M, Zhu W, Fu Y, Sun X. Community-based heat-sensitive moxibustion for primary hypertension: study protocol for a randomized controlled trial with patient-preference arms. Trials. 2022 Feb 16;23(1):154. doi: 10.1186/s13063-022-06092-4. PMID 35172871